CLINICAL TRIAL: NCT03453476
Title: Effect of Photodynamic Therapy on Gingival Crevicular Cytokines in Periodontitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Foo Lean Heong, Periodontic Resident, Faculty of Dentistry, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NUSingapore
Record Dates: First submitted 2018-01-23; First posted 2018-03-05 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-02

CONDITIONS: Periodontitis, Adult; Periodontal Pocket; Periodontitis; Periodontal Attachment Loss
Keywords: Photodynamic therapy; Interleukin 1-beta; Tumour necrosis factor - alpha; Interleukin-6; Interleukin-8; Matrix metalloproteinase-8
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Pocket; Periodontitis; Periodontal Attachment Loss

STUDY DESIGN:
Intervention Model Description: Split-mouth design
Who Masked: Participant, Care Provider, Investigator
Masking Description: Allocation of test and control quadrants were done randomly by asking each study participant to choose either numbers "1" or "2". Number "1" defined quadrants 1 and 3 as the test quadrants while number "2" referred to quadrants 2 and 4 as the test quadrants. The remaining quadrants served as the control quadrants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SRP and Fotosan 630 (Experimental): Scaling and root planing, photodynamic therapy using Fotosan 630
  Interventions: Device: SRP and Fotosan 630
- Control (No Intervention): Scaling and root planing only

INTERVENTIONS:
Device: SRP and Fotosan 630 — After isolating the test quadrants with cotton roll, toluidine blue was applied into the deep pockets (PD ≥ 4mm) at the test quadrants for 10 seconds, followed by inserting a perio tip (15 or 21 mm depending on the depth of the pocket) that connected to a LED emitting device, and light was emitted for 20 seconds. Toluidine blue in the deep pocket was removed by injecting normal saline into the pocket.
  Other Names: Fotosan 630, CMS Dental, Copenhagen, Denmark
  Arms: SRP and Fotosan 630

SUMMARY:
Systemically healthy periodontitis patients were recruited in this single-blind, split-mouth, randomized controlled clinical trial. After SRP, PDT was applied at probing depth (PD) ≥ 4 mm at test quadrant. At baseline, 3rd month and 6th month, clinical parameters and cytokine pattern in gingival crevicular fluids (GCFs) were analysed.

DETAILED DESCRIPTION:
Periodontal parameters and cytokine IL-1β, IL-6, IL-8, TNF-α, MMP-8 levels were analysed.

ELIGIBILITY:
Inclusion Criteria:

* Adults who were medically fit or have medical condition that did not alter the outcome of periodontal treatment.
* Females who were not pregnant or nursing.
* Controlled diabetes mellitus with HbA1c < 7.5 mmol/L.
* Not on any antibiotics or steroids 3 months prior to periodontal treatment.
* Diagnosed to have either localized or generalized chronic or aggressive periodontitis (Armitage, 1999) with all 4 quadrants having at least 2 sites with probing depth ≥ 4 mm.
* Consented to follow the non-surgical periodontal treatment (scaling and root planing) with PDT throughout the period of study, i.e. approximately 6 months.

Exclusion Criteria:

* Allergic to photosensitizer or dye
* Pregnant lady and nursing mothers
* Uncontrolled diabetes

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-03-31 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline probing depth at 3rd month and 6th month | 3 months and 6 months
  Clinical probing depth in mm
Changes from baseline clinical attachment level at 3rd month and 6th month | 3 months and 6 months
  Clinical attachment level in mm
Changes from baseline gingival recession level at 3rd month and 6th month | 3 months and 6 months
  Gingival recession level in mm
Changes from baseline bleeding score at 3rd month and 6th month | 3 months and 6 months
  Bleeding score in percentage
Changes from baseline Interleukin-1 level at 3rd month and 6th month | 3 months and 6 months
  Interleukin-1 level in gingival crevicular fluid
Changes from baseline Interleukin-6 level at 3rd month and 6th month | 3 months and 6 months
  Interlekin-6 level in gingival crevicular fluid
Changes from baseline Interleukin-8 level at 3rd month and 6th month | 3 months and 6 months
  Interleukin-8 level in gingival crevicular fluid
Changes from baseline Tumour necrosis factor-alpha level at 3rd month and 6th month | 3 months and 6 months
  Tumour necrosis factor-alpha level in gingival crevicular fluid
Changes from baseline Matrix metalloproteinase-8 level at 3rd month and 6th month | 3 months and 6 months
  Matrix metalloproteinase-8 level in gingival crevicular fluid

CONTACTS AND LOCATIONS:
Overall Officials: Lum Peng Lim, Study Director — Faculty of Dentistry, National University of Singapore

IPD SHARING:
Plan to Share IPD: No